CLINICAL TRIAL: NCT03789708
Title: Study of Some Pharmacological and Biochemical Effects of Gum Arabic Supplementation to Hemodilaysis Patients
Brief Title: Effects of Gum Arabic Supplementation in Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Khartoum (Other)
Collaborators: National Center for Kidney Diseases and Surgery (Unknown); Almughtaribeen University (Unknown)
Responsible Party: Principal Investigator, Sarra Elamin, Assistant Professor, University of Khartoum
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 016227
Record Dates: First submitted 2018-12-27; First posted 2018-12-31 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Gum Arabic

STUDY DESIGN:
Intervention Model Description: Randomized and controlled clinical trial with parallel design
Who Masked: Participant, Care Provider
Masking Description: The placebo and the Gum Arabic are provided to patients in similar unlabeled packages
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A (Experimental): Patients will receive 10 g of Gum Arabic supplementation daily for four weeks. Gum Arabic is provided in the form of easily soluble granules. Participants are asked to dissolve it in water or juice and drink it.
  Interventions: Dietary Supplement: Gum Arabic
- B (Placebo Comparator): Patients will receive 5 g of maltodextrin supplementation daily for four weeks. Maltodextrin is an easily digested polysacharide provided in the form of soluble whitish powder that has no taste or odor. Participants are asked to dissolve it in water or juice and drink it.
  Interventions: Other: Placebo
- C (Experimental): Patients will receive 20 g of Gum Arabic supplementation daily for four weeks
  Interventions: Dietary Supplement: Gum Arabic
- D (Experimental): Patients will receive 40 g of Gum Arabic supplementation daily for four weeks
  Interventions: Dietary Supplement: Gum Arabic

INTERVENTIONS:
Dietary Supplement: Gum Arabic — Instantly soluble granules of Gum Arabic; 100% Acacia Senegal
  Arms: A; C; D
Other: Placebo — Maltodextrin powder, easily soluble
  Arms: B

SUMMARY:
Gum Arabic is a naturally produced gummy exudate from Acacia Senegal tree. It's a complex polysaccharide with proven prebiotic properties. Through its effect on intestinal bacteria, it's expected to reduce systemic levels of toxic bacterial metabolites and reduce inflammatory markers.By increasing fecal bacteria mass it's also expected to reduce blood urea level. These changes are potentially beneficial to hemodialysis patients who suffer from disturbed intestinal flora and a chronic inflammatory status. The investigators hypothesize that supplementing the diet of hemodialysis patients with Gum Arabic for four weeks would reduce inflammatory markers, increase total anti-oxidant capacity and reduce blood urea concentration.

ELIGIBILITY:
Inclusion Criteria:

* Adult end-stage renal disease patients maintained on regular hemodialysis

Exclusion Criteria:

* Chronic liver disease
* Malignant condition
* Inflammatory bowel disease
* History of bowel resection
* Long term antibiotic therapy
* Pregnancy or lactation
* Current use of immunosuppressive medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Highly sensitive C-reactive protein (hs CRP) level | 4 weeks
  Change in serum level of highly sensitive C-reactive protein.
Total anti-oxidant capacity | 4 weeks
  Change in serum total anti-oxidant capacity
Blood urea level | 4 weeks
  Change in urea blood level

SECONDARY OUTCOMES:
Serum calcium | 4 weeks
  Change in serum calcium level
Serum phosphorus | 4 weeks
  Change in serum phosphorus level
Serum uric acid | 4 weeks
  Change in serum uric acid level

CONTACTS AND LOCATIONS:
Overall Officials: Sarra Elamin, MD, Principal Investigator — Consultant Nephrologist
Locations (1):
- Doctor Salma Center for Kidney Diseases, Khartoum, Sudan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cooper TE, Khalid R, Chan S, Craig JC, Hawley CM, Howell M, Johnson DW, Jaure A, Teixeira-Pinto A, Wong G. Synbiotics, prebiotics and probiotics for people with chronic kidney disease. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD013631. doi: 10.1002/14651858.CD013631.pub2. PMID 37870148